CLINICAL TRIAL: NCT07371845
Title: The Effect of Teach-Back Education Given to Mothers of Preterm Infants on Breastfeeding Success and Mother-Infant Bonding: A Randomized Controlled Trial
Brief Title: Effect of Teach-Back Education on Breastfeeding and Bonding in Mothers of Preterm Infants
Acronym: TEACH-PRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Devran ATALAY ÖZKILIÇ, Clinical Researcher, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ATATURKU-HF-DAÖ-02
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Premature; Breast Feeding; Mother-Child Relationship
Keywords: teach-back; preterm infant; breastfeeding success
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups: an experimental group and a control group.
Masking Description: Data collection tools will be collected by an interviewer independent of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-back Education Group (Experimental): Mothers receive teach-back education on breastfeeding and infant care.
  Interventions: Behavioral: Teach-Back Education
- Control Group (No Intervention): Mothers receive routine care without teach-back education.

INTERVENTIONS:
Behavioral: Teach-Back Education — A structured teach-back education program is provided to mothers of preterm infants to improve breastfeeding practices and enhance mother-infant bonding. Mothers are asked to repeat and demonstrate the information to confirm understanding.
  Arms: Teach-back Education Group

SUMMARY:
The aim of this randomized controlled experimental study is to contribute to the standardization of nursing interventions for premature mothers and to establish a scientific basis for breastfeeding education models in our country. It also aims to evaluate the effects of the following: digital privacy literacy, children's autonomy, decision-making ability, and privacy awareness. The hypotheses of the study are as follows:

H₁: Mothers who received Teach-Back training have a higher level of breastfeeding self-efficacy.

H₂: Mothers who received Teach-Back training have a higher level of mother-infant bonding.

H₀: There is no significant difference between the groups.

DETAILED DESCRIPTION:
The study will be conducted with mothers of premature babies who meet the inclusion criteria at the state hospital located in Tatvan district, affiliated with the Bitlis Provincial Health Directorate. Participants will be assigned to two groups using simple random sampling:

1. Experimental group: (Mothers who received Teach-Back training)
2. Control group: (Mothers who received routine discharge education). Data will be collected using the "Participant Identification Form", "Breastfeeding Self-Efficacy Scale for Mothers of Preterm Babies", "Mother-Infant Bonding Scale" and "Teach-Back Training Evaluation Form".

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Having a baby born before the 37th week of gestation (being a mother of a premature baby),
* Being able to read and understand Turkish,
* Having actually started breastfeeding,
* Having no hearing, visual, or cognitive communication impairment,
* Not having a diagnosed serious psychiatric illness (major depression, anxiety disorder, etc.),
* The baby not being in a serious clinical condition, not under palliative care or intensive life support,
* Not participating in another breastfeeding education or counseling program at the same time,
* Voluntarily agreeing to participate in the study.

Exclusion Criteria:

* All mothers who do not meet the inclusion criteria will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — prematüre bebek anneleri
Enrollment: 102 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Participant Introduction Form | First week
  The form was prepared by the researcher in accordance with the literature to determine the sociodemographic (age, education level, income level, marital status, place of residence) and obstetric characteristics (number of pregnancies, mode of delivery, gestational age, birth weight, neonatal hospital stay, previous breastfeeding experience, etc.) of the mothers participating in the study. The form was developed using research examining the relationships between breastfeeding self-efficacy, mother-infant bonding, and maternal characteristics.
The Breastfeeding Self-Efficacy Scale for Mothers of Ill and/or Preterm Infants | First Week
  This scale was developed by Wheeler and Dennis (2013) and adapted into Turkish by Aluş Tokat et al. (2020). It is an 18-item scale with a 5-point Likert scale (1=Not sure at all, 2=Not sure at all, 3=Sometimes sure, 4= Sure, 5=Very sure). The minimum score obtainable on the scale is 18, and the maximum is 90. A higher score indicates high breastfeeding self-efficacy.
Mother-to-Infant Bonding Scale | First Week
  This scale was developed by Taylor et al. (2005), and its Turkish validity and reliability study was conducted by Aydemir-Karakulak (2009). The scale consists of 8 items. It uses a 4-point Likert scale (1 = none - 4 = very much). Scores on the scale range from 0 to 24. The Cronbach alpha coefficient was found to be 0.683.

SECONDARY OUTCOMES:
The Breastfeeding Self-Efficacy Scale for Mothers of Ill and/or Preterm Infants | within the fist week
  This scale was developed by Wheeler and Dennis (2013) and adapted into Turkish by Aluş Tokat et al. (2020). It is an 18-item scale with a 5-point Likert scale (1=Not sure at all, 2=Not sure at all, 3=Sometimes sure, 4= Sure, 5=Very sure). The minimum score obtainable on the scale is 18, and the maximum is 90. A higher score indicates high breastfeeding self-efficacy.
Mother-to-Infant Bonding Scale | within the first week
  This scale was developed by Taylor et al. (2005), and its Turkish validity and reliability study was conducted by Aydemir-Karakulak (2009). The scale consists of 8 items. It uses a 4-point Likert scale (1 = none - 4 = very much). Scores on the scale range from 0 to 24. The Cronbach alpha coefficient was found to be 0.683.
Teach-Back Training Evaluation Form | within the first week
  This form was prepared by the researcher to observe the comprehensibility and learning level of the Teach-back training given to the experimental group. The form evaluates the participant's ability to explain the information received in their own words, recall basic concepts, and express their application plan. A short checklist consisting of five items is completed observationally at the end of each session with a score of 0-2 (insufficient-partially sufficient). The form will only be used to monitor the quality of the training process. This evaluation approach is consistent with international guidelines for monitoring the process accuracy of the teach-back method.

CONTACTS AND LOCATIONS:
Overall Officials: fatma güdücü tüfekci, Study Director — Ataturk University
Locations (1):
- Atatürk Üniversitesi, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No